CLINICAL TRIAL: NCT01196611
Title: Effectiveness of Two Therapeutic Approaches in Female Teachers With Voice Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Leticia Caldas Teixeira, Professor/PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETIC 0521.0.203.000-09
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2010-09

CONDITIONS: Voice Disorders
Keywords: Voice disorders; Voice
MeSH Terms: conditions — Voice Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Function Voice Exercises (Experimental): Behavioral: Function Voice Exercises Patients will receive 6 sessions of therapy over a course of 6 weeks, with one session per week.
  Interventions: Behavioral: Function Voice Exercises
- Voice amplification (Experimental): Behavioral: Voice amplification Patients will use VA over a course of 6 weeks.
  Interventions: Behavioral: Voice Amplification

INTERVENTIONS:
Behavioral: Voice Amplification — Behavioral: Voice Amplification. Patients use VA over a course of 6 weeks Control group. No treatment over a course of 6 weeks.
  Arms: Voice amplification
Behavioral: Function Voice Exercises — Function Voice Exercises Patients will receive 6 sessions of therapy over a course of 6 weeks, with one session per week.
  Arms: Function Voice Exercises

SUMMARY:
The study compares two different approaches of voice therapy. Vocal Functional Exercises (Stemple,1997) and Voice Amplification using a portable amplifier (Tsi Supervoz II - Tecnisystem do Brasil TSI 1210).

DETAILED DESCRIPTION:
Both approaches combined with Vocal Hygiene Program (Behlau, 2007).The target population are female teachers because they have the highest risk for developing voice problems. For this study the investigators are primarily interested in seeing if Vocal Functional Exercises and Voice Amplification are equally effective at improving vocal functioning in teachers with voice disorders. The Fiberoptic endoscopic evaluation will be done before randomization. All the participants will complete before and after a 6-week treatment phase (a) Voice Activity and Participation Profile (PPAV), an instrument designed to appraise the self-perceived psychosocial consequences of voice disorders to assess the impact of voice disorders on daily activities (b) Audio voice recording for later acoustic analysis, through the Kay Elemetrics Multi Dimensional Voice Program (c) Audio recording for later perceptual analysis through Consensus Auditory-Perceptual Evaluation of Voice (CAPE_V). It is believed that the search for evidence in clinical studies like this can contribute to awareness programs and vocal training for teachers.

ELIGIBILITY:
Inclusion Criteria:

* Female teacher
* 21-50 years old.
* Full or part time elementary to middle school teacher ( Prefeitura Municipal de Belo Horizonte).
* Minimum 20 hour weekly workload.
* Medical reference to speech therapy due to behavioral dysphonia

Exclusion Criteria:

* Physical education or daycare teachers.
* Professional singers.
* Neurological and/or psychiatric voice disorders

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Fiberoptic endoscopic evaluation | One year
Score(CAPE_V); score(PPAV); score on acoustic analysis | One year

CONTACTS AND LOCATIONS:
Overall Officials: Mara S Behlau, PhD, Study Director — Universidade Federal de São Paulo; Arnaldo L Colombo, PhD, Study Director — Federal University of São Paulo; Letícia C Teixeira, MsC, Principal Investigator — Federal University of São Paulo; Ana Cristina C Gama, D, Study Director — Federal University of Minas Gerais
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The data of the participants are confidential